CLINICAL TRIAL: NCT05793775
Title: Circulating Tumor Cells and Neutrophils Count for Colorectal Metastatic Cancer
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 10-AOI-05
Record Dates: First submitted 2012-03-23; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2012-01

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples

SUMMARY:
Colorectal cancer represents a major public health problem in France because of its high incidence and severe prognosis. Early stages of the disease are well know and have justified the establishment of a mass screening strategy. Unfortunately, the factors determining the progression to metastatic disease about them much harder to grasp. Various prognostic factors and predictors of treatment response have been identified and are being used but most of them are In practice, they are sometimes coarse and relatively little discriminant for patients.

It is now possible to directly quantify the amount of circulating tumor cells in peripheral blood. Quantification of circulating tumor cells beyond a threshold of 3 cells/7,5 ml has been established as a major prognostic factor, and the rapid decrease in the number of these cells under treatment is also a predictor of response for patients suffering from metastatic colorectal cancer . Furthermore, it has also been shown that the quality and importance of the systemic and peritumoral inflammatory response in carcinomas, including colorectal, played a key role in the prognosis of patients. In particular, the presence of high levels of blood neutrophils has been raised by many studies as being followed by a poorer prognosis.

However, the correlation between the presence of circulating tumor cells and high levels of neutrophils has never been studied. There is a rational to assume that this association exists, and secondly that the presence of circulating tumor cells in a proinflammatory environment represented by a high levels of blood neutrophils promotes metastasis by exerting a negative synergistic effect on the prognosis of patients.

The main objective of this pilot study is to find a correlation between the amount of circulating neutrophils and the presence of circulating tumor cells in patients with colon cancer metastatic unresectable non-pretreated. The secondary objective is to investigate whether this association results in a negative synergistic effect in terms of progression-free survival and survival to one year. This is a non-interventional study. The investigators expect the inclusion in one year of thirty patients in two centers (University Hospital Centre Antoine Lacassagne Nice) to achieve these goals.

ELIGIBILITY:
* Inclusion criteria:

  * Age > 18 years
  * Metastatic colorectal cancer
  * Chemotherapy required
  * Measurable scannographic target
  * CT-scan < 3 weeks
  * Written consent

Non-inclusion criteria :

* Personal history of invasive carcinoma
* Prior chemotherapy regimen
* Treatment with G-CSF analogs
* Corticotherapy

Exclusion criteria:

• Consent withdrawal

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Research of an association between polymorphonuclear count (number of cells per liter) and circulating tumor cells number (number of circulating tumor cells per 7,5 mililiters. | one time

SECONDARY OUTCOMES:
Research of a synergistic effect between high polymorphonuclear count and high level of circulating tumor cells on progression-free survival and overall survival. Progression will be defined according to RECIST criteria. | one time

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Gastroentérologie et de Nutrition - CHU de Nice - Hôpital de l'Archet, 151 route de Saint-Antoine de Ginestière, Nice
  - Département d'Oncologie médicale - Centre Antoine Lacassagne, Nice